CLINICAL TRIAL: NCT00058318
Title: A Phase II Study of IV Gemcitabine and Oral Capecitabine in Patients With Advanced Renal Cell Cancer
Brief Title: S0312, Gemcitabine and Capecitabine in Treating Patients With Advanced Renal Cell (Kidney) Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000288820; U10CA032102 (NIH); S0312 (Other: SWOG)
Record Dates: First submitted 2003-04-07; First posted 2003-04-09 (Estimated); Last update posted 2012-11-02 (Estimated); Status verified 2012-10

CONDITIONS: Kidney Cancer
Keywords: stage IV renal cell cancer; stage III renal cell cancer
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell | interventions — Capecitabine; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Experimental): Gemcitabine + Capecitabine
  Interventions: Drug: capecitabine; Drug: gemcitabine hydrochloride

INTERVENTIONS:
Drug: capecitabine — Capecitabine will be given 625 mg/m^2 (1250 mg/m^2/day) by mouth twice a day on day 1-21 for every cycle (1 cycle =28 days) until disease progression
Drug: gemcitabine hydrochloride — Gemcitabine will be given 900 mg/m^2 by intravenous infusion over 30 minutes on day 1, 8, and 15 for every cycle (1 cycle = 28 days) until disease progression.

SUMMARY:
RATIONALE: Drugs used in chemotherapy such as gemcitabine and capecitabine use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one chemotherapy drug may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combining gemcitabine with capecitabine in treating patients who have advanced renal cell cancer (kidney cancer).

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine response (confirmed and unconfirmed complete and partial) of patients with advanced renal cell cancer treated with gemcitabine and capecitabine.
* Determine the 6-month time to treatment failure rate and overall survival rate of patients treated with this regimen.
* Determine the qualitative and quantitative toxic effects of this regimen in these patients.
* Correlate, preliminarily, tumor response with the intratumoral content of the enzymes involved in the activation and degradation of these drugs in these patients.

OUTLINE: Patients receive gemcitabine IV over 30 minutes on days 1, 8, and 15 and oral capecitabine twice daily on days 1-21. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months for 1 year and then every 6 months for 2 years.

PROJECTED ACCRUAL: A total of 38 patients will be accrued for this study within 3.8-4.2 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed renal cell carcinoma

  * Metastatic (M1) disease OR
  * M0 provided the primary tumor is unresectable
* Measurable disease

  * At least 1 unidimensionally measurable lesion
  * Soft tissue disease that has been irradiated within the past 2 months is not considered measurable disease
  * Soft tissue disease within a prior radiation field is measurable provided it has progressed since therapy and there is also measurable disease outside of the irradiated field
* No prior or concurrent brain metastases

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Zubrod 0-2

Life expectancy

* Not specified

Hematopoietic

* Absolute granulocyte count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* Aspartate aminotransferase (SGOT) no greater than 1.5 times ULN

Renal

* Creatinine clearance at least 50 mL/min

Cardiovascular

* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia

Other

* Not pregnant or nursing
* Fertile patients must use effective contraception
* No other concurrent uncontrolled illness that would preclude study participation
* No psychiatric illness or social situation that would preclude study compliance
* No uncontrolled diabetes mellitus
* No ongoing or active infection
* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer, carcinoma in situ of the cervix, or stage I or II cancer currently in complete remission

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No more than 2 prior immunotherapy regimens comprising interferon (IFN) and/or interleukin-2 (IL-2)
* At least 28 days since prior IFN or IL-2 and recovered

Chemotherapy

* No prior chemotherapy for renal cell cancer

Endocrine therapy

* Not specified

Radiotherapy

* See Disease Characteristics
* No prior radiotherapy to 25% or more of the bone marrow
* At least 21 days since prior radiotherapy and recovered

Surgery

* At least 28 days since prior surgery and recovered
* Prior resection of the primary tumor allowed (in patients with metastatic disease)

Other

* At least 4 weeks since prior sorivudine or brivudine
* No concurrent sorivudine or chemically related analogues (e.g., brivudine)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2004-12; Primary Completion 2007-05 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Response | every 8 weeks until progression

SECONDARY OUTCOMES:
Survival | every 8 weeks while on treatment, then every 3 months for first year, then every 6 months for 3 years
Time to treatment failure | every 8 weeks until progression

CONTACTS AND LOCATIONS:
Overall Officials: Peter J. VanVeldhuizen, MD, Study Chair — Kansas City Veteran Affairs Medical Center

REFERENCES:
- [Result] Van Veldhuizen PJ, Hussey M, Lara PN Jr, Mack PC, Gandour-Edwards R, Clark JI, Lange MK, Crawford DE. A phase ii study of gemcitabine and capecitabine in patients with advanced renal cell cancer: Southwest Oncology Group Study S0312. Am J Clin Oncol. 2009 Oct;32(5):453-9. doi: 10.1097/COC.0b013e3181925176. PMID 19487915
- [Result] van Veldhuizen PJ, Hussey M, Lara PN, et al.: A phase II study of IV gemcitabine (G) and oral capecitabine (C) in patients (pts) with advanced renal cell cancer (RCC): results of Southwest Oncology Group study 0312. [Abstract] J Clin Oncol 25 (Suppl 18): A-15562, 654s, 2007.